CLINICAL TRIAL: NCT05887778
Title: Effect of Systematic Dexamethasone on the Duration of Supraclavicular Brachial Plexus Block for Anesthesia After Pediatric Hand/Wrist Surgery
Brief Title: Dexamethasone in Supraclavicular Brachial Plexus Block for Anesthesia After Pediatric Hand/Wrist Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9/2023
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Wrist Disease; Hand Injuries and Disorders
MeSH Terms: conditions — Hand Injuries; Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo injection (Active Comparator): 5ml of 0,9% sodium chloride - before the popliteal nerve block
  Interventions: Drug: Sodium Chloride 0.9% Inj
- 0,1mg/kg Dexamethasone (Active Comparator): 0,1mg/kg dexamethasone sodium phosphate - before the popliteal nerve block
  Interventions: Drug: 0,1mg/kg Dexamethasone
- 0,2 mg/kg Dexamethasone (Active Comparator): 0,2 mg/kg dexamethasone sodium phosphate - before the popliteal nerve block
  Interventions: Drug: 0,2mg/kg Dexamethasone

INTERVENTIONS:
Drug: Sodium Chloride 0.9% Inj — administration of 5ml 0,9% sodium chloride - 30 minutes before the supraclavicular brachial plexus block
  Other Names: placebo
  Arms: placebo injection
Drug: 0,1mg/kg Dexamethasone — administration of 0,1mg/kg Dexamethasone - 30 minutes before the supraclavicular brachial plexus block
  Other Names: small dose
  Arms: 0,1mg/kg Dexamethasone
Drug: 0,2mg/kg Dexamethasone — administration of 0,2mg/kg Dexamethasone - 30 minutes before the supraclavicular brachial plexus block
  Other Names: large dose
  Arms: 0,2 mg/kg Dexamethasone

SUMMARY:
Effect of Systematic Dexamethasone on the Duration of Supraclavicular Brachial Plexus Block for Anesthesia After Pediatric Hand/Wrist Surgery

DETAILED DESCRIPTION:
This study is proposed to explore the effect of systemic Dexamethasone on the duration of supraclavicular brachial plexus block for analgesia after pediatric ankle surgery.

After hand and wrist surgery, children need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anesthesia is essential in children due to the much lower toxicity threshold of local anesthetics. An effective adjuvant, such as Dexamethasone, could allow for a higher dilution of local anesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone use has been compared in adults. However, there is a massive lack of research regarding children.

In this study, investigators compare different doses of systemic Dexamethasone. Before the anesthesia, the patients receive Dexamethasone intravenously. Groups 2 and 3 have dexamethasone doses of 0.1mg/kg and 0.2mg/kg.

The investigator's goal is to find a dexamethasone dose that is as low as possible but simultaneously covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for hand/wrist surgery
* body weight > 5kg

Exclusion Criteria:

* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid Consumption | 48 hours
  Total opiate consumption after surgery
Pain score | 4 hours, 8 hours, 12 hours, 16 hours, 18 hours, 24 hours, 28 hours, 32 hours, 36 hours, 40 hours, 44 hours, 48 hours after surgery
  children <3years old FLACC score (Face, Legs, Activity, Cry, Consolability) children >3years old NRS (Numerical Rating Scale)
Blood glucose | 24 and 48 hours after surgery
  Blood glucose every 24 hour during hospitalization
NLR | 24 and 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 24 and 48 hours after surgery
  Platelet-to-lymphocyte ratio
Mobilisation | 4 hours, 8 hours, 12 hours, 16 hours, 18 hours, 24 hours, 28 hours, 32 hours, 36 hours, 40 hours, 44 hours, 48 hours after surgery
  Finger movement every 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Romanowski, Prof.dr hab, Study Director — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided